CLINICAL TRIAL: NCT06593548
Title: A Prospective, Single-arm, Single-center, Phase II Clinical Study of Ivosidenib (AK112) Combined With CapeOX and Radiotherapy in Patients With Unresectable Metastatic MSS-type Colorectal Cancer: Efficacy and Safety Assessment
Brief Title: Lvosidenib (AK112) Combined With CapeOX and Radiotherapy in Patients With Unresectable Metastatic MSS-type Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, LI XIN-XIANG, professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Miracle-03
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: CRC; MSS; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — ivosidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- AK112 combined with CapeOX and radiotherapy (Experimental): Participants will receive Ivosidenib in combination with CapeOX chemotherapy and radiotherapy. Participants will first receive Ivosidenib in combination with CapeOX during the first cycle, followed by radiotherapy starting 2 weeks after medication.
  Interventions: Drug: Ivosidenib (AK112)

INTERVENTIONS:
Drug: Ivosidenib (AK112) — Participants will receive Ivosidenib in combination with CapeOX chemotherapy and radiotherapy. Participants will first receive Ivosidenib in combination with CapeOX during the first cycle, followed by radiotherapy starting 2 weeks after medication. Depending on the dose limits of normal tissue radiation, Stereotactic Ablative Radiotherapy (SABR), large fraction radiotherapy, or high-dose combined with low-dose radiotherapy will be administered to primary and metastatic lesions. One week after completing radiotherapy, participants will continue to receive Ivosidenib in combination with CapeOX systemic treatment. If primary and metastatic lesions are too extensive for initial radiotherapy, participants will continue to receive Ivosidenib in combination with CapeOX systemic treatment until the lesions shrink, at which point radiotherapy may be considered.。

SUMMARY:
This is a prospective, single-arm, single-center Phase II clinical study. In this study, participants will receive Ivosidenib in combination with CapeOX chemotherapy and radiotherapy. The treatment regimen is as follows: participants will first receive Ivosidenib in combination with CapeOX chemotherapy during the first cycle, followed by radiotherapy starting 2 weeks after medication. Depending on the dose limits of normal tissue radiation, Stereotactic Ablative Radiotherapy (SABR), large fraction radiotherapy, or high-dose combined with low-dose radiotherapy will be administered to primary and metastatic lesions. One week after completing radiotherapy, participants will continue to receive Ivosidenib in combination with CapeOX systemic treatment. If extensive primary and metastatic lesions cannot be treated with radiotherapy initially, participants will continue to receive Ivosidenib in combination with CapeOX systemic treatment until the lesions shrink, at which point radiotherapy may be considered.

Assessments will be conducted every 2 treatment cycles after treatment initiation, with multidisciplinary team (MDT) discussions to determine if No Evidence of Disease (NED) is achieved. Patients achieving NED may undergo surgery or local treatment, while those with stable or partial responses will continue combination therapy. Patients with disease progression will discontinue study treatment. Patients ineligible for surgical treatment will continue combination therapy until disease progression or until they exit the study for surgical treatment.

During the study period, participants will undergo safety monitoring. The safety follow-up period is defined as 90 days after the last dose of Ivosidenib. Safety data will be collected from the time of informed consent signing until the end of the safety follow-up period or initiation of new anti-tumor treatment (whichever occurs first).

DETAILED DESCRIPTION:
This is a prospective, single-arm, single-center Phase II clinical study. In this study, participants will receive Ivosidenib in combination with CapeOX chemotherapy and radiotherapy. The treatment regimen is as follows: participants will first receive Ivosidenib in combination with CapeOX chemotherapy during the first cycle, followed by radiotherapy starting 2 weeks after medication. Depending on the dose limits of normal tissue radiation, Stereotactic Ablative Radiotherapy (SABR), large fraction radiotherapy, or high-dose combined with low-dose radiotherapy will be administered to primary and metastatic lesions. One week after completing radiotherapy, participants will continue to receive Ivosidenib in combination with CapeOX systemic treatment. If extensive primary and metastatic lesions cannot be treated with radiotherapy initially, participants will continue to receive Ivosidenib in combination with CapeOX systemic treatment until the lesions shrink, at which point radiotherapy may be considered.

Assessments will be conducted every 2 treatment cycles after treatment initiation, with multidisciplinary team (MDT) discussions to determine if No Evidence of Disease (NED) is achieved. Patients achieving NED may undergo surgery or local treatment, while those with stable or partial responses will continue combination therapy. Patients with disease progression will discontinue study treatment. Patients ineligible for surgical treatment will continue combination therapy until disease progression or until they exit the study for surgical treatment.

During the study period, participants will undergo safety monitoring. The safety follow-up period is defined as 90 days after the last dose of Ivosidenib. Safety data will be collected from the time of informed consent signing until the end of the safety follow-up period or initiation of new anti-tumor treatment (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75.
* ECOG performance status of 0-1.
* Initial diagnosis confirmed by colonoscopy and pathology as colorectal adenocarcinoma.
* Imaging confirmation of multiple measurable metastases, deemed unresectable initially after MDT discussion.
* No prior treatment or more than 1 year since completion of initial untreated/post-operative adjuvant chemotherapy, and no previous anti-tumor therapy thereafter.
* With good organ function, without contraindications for surgery or chemotherapy.
* Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN, and international normalized ratio (INR) ≤ 1.5 × ULN (if not receiving anticoagulant therapy).
* Urine protein < 2+; if urine protein ≥ 2+, 24-hour urine protein quantitative test must show ≤ 1g protein.
* Left ventricular ejection fraction (LVEF) ≥ 55%. 12-lead electrocardiogram: Fridericia-corrected QT interval (QTcF) < 470 msec.
* Expected survival > 6 months.
* Clear status of KRAS, NRAS, BRAF, and HER2 genes.
* Microsatellite stable or mismatch repair protein proficient patients.

Exclusion Criteria:

* Age <18 years or >75 years.
* History of any other malignancy within 5 years, except adequately treated cervical carcinoma in situ, squamous cell carcinoma of the skin, or basal cell carcinoma that has been effectively controlled.
* Malignant pleural or peritoneal effusion.
* Severe internal medical complications preventing chemotherapy or surgery.
* Clinical or radiological evidence of spinal cord compression, or tumor within 3 mm of the spinal cord on MRI.
* Imaging-confirmed brain, ovarian, or peritoneal metastases.
* Patients deemed suitable for aggressive systemic treatment to achieve conversion after MDT discussion.
* Pathologically diagnosed signet ring cell carcinoma.
* Patients with microsatellite instability or mismatch repair protein deficiencies.
* Patients with intestinal obstruction, perforation, bleeding requiring emergency surgical resection.
* Immunodeficiency diseases, including primary immunodeficiency diseases (genetically determined) or secondary immunodeficiency diseases.
* Known or suspected interstitial pneumonia.
* Severe cardiovascular diseases, including but not limited to conditions meeting NYHA class (III or higher), myocardial infarction or cerebrovascular accident (ischemic stroke, symptomatic cerebral infarction) within the past 3 months prior to first dosing, unstable angina or unstable arrhythmias within the past 1 month prior to first dosing, congestive heart failure beyond the above criteria, symptomatic superior vena cava syndrome, etc.
* Venous thromboembolic events within the past 3 months, such as deep vein thrombosis and pulmonary embolism.
* History of receiving live attenuated vaccines within 28 days prior to first study drug administration or anticipated need for live attenuated vaccines during the study period.
* Active hepatitis B (defined as positive hepatitis B surface antigen [HBsAg] with HBV-DNA ≥500 IU/ml).
* Hepatitis C (defined as positive hepatitis C virus antibody [HCV-Ab]).
* History of tuberculosis infection or treatment within the past 1 year prior to signing informed consent.
* History of or planned allogeneic bone marrow or solid organ transplantation.
* Abnormal coagulation function (INR > 1.5 or APTT > 1.5 × ULN), with bleeding tendency or undergoing thrombolysis or requiring long-term anticoagulant therapy with warfarin or heparin, or requiring long-term antiplatelet therapy (aspirin ≥ 300 mg/day or clopidogrel ≥ 75 mg/day).
* Peripheral neuropathy of Grade ≥2 according to NCI-CTCAE v5.0.
* Concurrent other infectious diseases unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
PFS | The time from the start of treatment until disease progression (PD) or death from any cause，whichever came first, assessed up to 100 months
  Progression-Free Survival (PFS)

CONTACTS AND LOCATIONS:
Locations (1):
- Xinxiang Li, Shanghai, Shanghai Municipality, China